CLINICAL TRIAL: NCT05951452
Title: The Developmental Origins of Endometriosis
Acronym: ENDOHaD
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other); Fondation pour la Recherche sur l'Endométriose (Unknown); Fondation pour la Recherche Médicale (Other); Université Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL23_0057
Record Dates: First submitted 2023-06-29; First posted 2023-07-19 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Endometriosis
Keywords: Endometriosis; Testosterone; Oxytocin; DOHaD
MeSH Terms: conditions — Endometriosis; Developmental Origins of Health and Disease | interventions — Blood Specimen Collection; Testosterone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serums and saliva extracts before and after wathching the empathy-inducing video
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ENDO +: Patients with endometriosis diagnosed by Magnetic Resonance Imaging (MRI) or laparoscopy
  Interventions: Other: Blood samples for testosterone and SHBG measurements; Other: Saliva samples for oxytocin measurements
- ENDO -: Patients without endometriosis diagnosed by laparoscopy
  Interventions: Other: Blood samples for testosterone and SHBG measurements; Other: Saliva samples for oxytocin measurements

INTERVENTIONS:
Other: Blood samples for testosterone and SHBG measurements — Several measurements of the testosterone concentration will be performed on serum from 10 mL of blood collected at:
  * t0 corresponding to the start of the hospital appointment and before watching the video
  * t1 which corresponds to 20 minutes after watching a 2 minutes empathy-inducing video
Other: Saliva samples for oxytocin measurements — Several measurements of the oxytocin concentration will be performed on 2 ml saliva samples:
  * t0 corresponding to 20 minutes after the start of the hospital appointment and before watching the video
  * t1 which corresponds to 20 minutes after watching a 2 minutes empathy-inducing video

SUMMARY:
Introduction:

Endometriosis is a common pathology affecting one in 10 women, characterized by the ectopic development of endometrium, which can cause pain and/or infertility. This pathology is primarily determined by hereditary factors, but it is also susceptible to environmental influences, such as the age of the onset of menstruation or exposure to chemical substances that modify the endocrine system. Recent studies have highlighted that endometriosis is more common in women with relatively short ano-genital distances (AGD), and that sensitivity to pain is closely linked to adult levels of testosterone (T) or oxytocin (OT).

Aim:

The main objective is to compare the anogenital distance (AGD) between two groups of women: one with stage III or IV endometriosis (ENDO +) and another group without endometriosis confirmed by laparoscopy (ENDO -).

The secondary objectives are to compare various factors between the 2 groups :

* Basal testosterone levels in blood.
* Variations in blood testosterone levels before and after a video stimulating empathy.
* Basal oxytocin levels in saliva.
* Variations in oxytocin levels in saliva before and after an empathy-stimulating video.
* Pelvic pain, between D2 and D5 after the start of the menstrual cycle.

For the ENDO + group only:

* Evaluate patients' quality of life, between D2 and D5 after the start of the menstrual cycle.
* Correlate pain experienced over the last 4 weeks with hormonal markers (AGD, T, OT).

Methods:

Participants in the ENDO+ group will fill in a questionnaire assessing the impact of pain experienced over the past 4 weeks on their quality of life. D0 is defined as the day when participants experience a menstrual bleed before 10 am. All participants will return for project-specific hospital appointment between D2 and D5 after the start of their menstrual cycle to measure T, Sex Hormone-Binding Globulin (SHBG) and OT.

During this consultation, the following samples will be taken:

* 10mL blood sample
* 2mL saliva sample

Both samples will be taken at t0 (before watching the video) and t1 (20 minutes after watching the video).

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous woman
* No hormonal contraception for at least 3 months
* Regular menstrual cycles (between 26 and 32 days) or proven ovulation (positive urine ovulation test ovulation test or progesterone level >3 ng/ml in the luteal phase)
* Normal BMI (≥ 18,5 and < 30 kg/m²)

Specific criteria (ENDO+ group) :

* Stage III or IV endometriosis confirmed by laparoscopy or by laparotomy or MRI
* Painful symptoms

Specific criteria (ENDO- group) :

• Patient without endometriosis confirmed by laparoscopy

Exclusion Criteria:

* Ovarian stimulation planned within 3 months
* Adenomyosis
* Use of a copper coil
* Polycystic ovary syndrome
* Pudendal neuralgia
* Episiotomy or lesion of the posterior perineum that may modify AGD
* Diabetes or thyroid disease
* Chronic liver failure, chronic renal failure, cardiac pathology, autoimmune disease
* Autism
* Diagnosis and/or treatment for psychiatric illness
* Chronic exposure to cocaine, methamphetamine, morphine or ecstasy within 30 days before the inclusion visit
* Chronic exposure to Tetrahydrocannabinol (THC) within 7 days prior to inclusion.
* Patient on treatment(s) that vary oxytocin (e.g. atosiban), testosterone or GnRH
* Pregnant or breast-feeding patient
* Patients who have given birth or breastfed within 6 weeks before the inclusion visit
* Patient unable to read French
* Failure to obtain informed consent
* Patient not affiliated with or not benefiting from a national health insurance scheme
* Person under legal protection, guardianship or curatorship
* Patient participating in other research involving the human person

Ages: 20 Years to 38 Years | Sex: Female
Age Groups: Adult
Study Population: Women with or without endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-01-08 (Estimated); Study Completion 2026-01-08 (Estimated)

PRIMARY OUTCOMES:
Measure of the anogenital distance (AGD) | At diagnosis or at inclusion
  AGD is measured at enrollment for patients already diagnosed by Magnetic resonance imaging (MRI), and it is measured during the laparoscopy once the diagnosis has been confirmed.
  AGD is measured by 2 different operators with a millimetric precision ruler according 2 validated methods :
  * measure of the distance from the clitoral surface to the anus (AGD-AC), and
  * measure of the distance from the posterior fourchette to the anus (AGD-AF). The method is described here: https://www.jove.com/v/57912/ Each operator will measure the AGD-AC and the AGD-AF 3 times. For each type of AGD, the final value will correspond to the mean of the 6 values.

SECONDARY OUTCOMES:
Basal total testosterone | t0 : Between the second and the fifth day of the menstrual cycle, before wathching an empathy-inducing video
  The basal total testosterone (Ttotal(t0)) level is measured in blood
Basal bio-available testosterone | t0 : Between the second and the fifth day of the menstrual cycle, before wathching an empathy-inducing video
  The basal bio-available testosterone (Tbio-available(t0)) level is measured in blood
Basal sex hormone-binding globulin | t0 : Between the second and the fifth day of the menstrual cycle, before watching an empathy-inducing video
  Basal sex hormone-binding globulin (SHBG(t0)) level is mesured in blood
Basal Free Androgen Index | t0 : Between the second and the fifth day of the menstrual cycle, before watching an empathy-inducing video
  Basal Free Androgen Index (FAI(t0)) = (Ttotal(t0)/SHBG(t0))*100
Total testosterone after empathy induction | t1 : Between the second and the fifth day of the menstrual cycle, after wathching an empathy-inducing video
  The total testosterone level after empathy induction (Ttotal(t1)) is measured in blood
Bio-available testosterone after empathy induction | t1 : Between the second and the fifth day of the menstrual cycle, after wathching an empathy-inducing video
  The bio-available testosterone level after empathy induction (Tbio-available(t1)) is measured in blood
Sex hormone-binding globulin after empathy induction | t1 : Between the second and the fifth day of the menstrual cycle, after wathching an empathy-inducing video
  Sex hormone-binding globulin after empathy induction (SHBG(t1)) is mesured in blood
Free Androgen Index after empathy induction | t1 : Between the second and the fifth day of the menstrual cycle, after wathching an empathy-inducing video
  Free Androgen Index after empathy induction (FAI(t1)) = (Ttotal(t1)/SHBG(t1))*100
Variation in total testosterone levels before and after an empathy-inducing video | t1 : Between the second and the fifth day of the menstrual cycle, after wathching an empathy-inducing video
  The level of variation in total testosterone before (t0) and after watching empathy-inducing video (t1) is assessed according to: Ttotal(t1)-Ttotal(t0)
Variation in bio-available testosterone levels before and after an empathy-inducing video | t1 : Between the second and the fifth day of the menstrual cycle, after wathching an empathy-inducing video
  The level of variation in bio-available testosterone before (t0) and after watching empathy-inducing video (t1) is assessed according to: Tbio-available(t1)-Tbio-available(t0)
Variation in Sex hormone-binding globulin levels before and after an empathy-inducing video | t1 : Between the second and the fifth day of the menstrual cycle, after wathching an empathy-inducing video
  The level of variation in Sex hormone-binding globulin before (t0) and after watching empathy-inducing video (t1) is assessed according to: SHBG(t1)-SHBG(t0)
% of variation in Free Androgen Index before and after an empathy-inducing video | t1 : Between the second and the fifth day of the menstrual cycle, after wathching an empathy-inducing video
  % of variation in Free Androgen Index before (t0) and after watching empathy-inducing video (t1) is assessed according to: [[FAI(t1)-FAI(t0)]/FAI(t0)] × 100
Basal oxytocin (OT) level | t0 : Between the second and the fifth day of the menstrual cycle, before wathching an empathy-inducing video
  The basal OT level is measured by the dosage in the saliva of :
  Total OT (OTtotal(t0))
Oxytocin (OT) level after empathy induction | t1 : Between the second and the fifth day of the menstrual cycle, after wathching an empathy-inducing video
  The basal OT level is measured by the dosage in the saliva of :
  Total OT (OTtotal(t1))
Variation in oxytocin (OT) level before and after an empathy-inducing video | t1 : Between the second and the fifth day of the menstrual cycle, after wathching empathy-inducing video
  Variation in OT level before (t0) and after watching an empathy-inducing video (t1) is assessed in the saliva according to:
  - OTtotal(t1)-OTtotal(t0)
  -% of variation of OT = [[OT(t1)-OT(t0)]/OT(t0)] × 100
Area under the Receiving Operator Characteristic (ROC) curve for AGD | At diagnosis (ENDO+) or at enrollment (ENDO-)
  The ROC curve is a graphical representation that illustrates the performance of a binary classification model. It plots the true positive rate (sensitivity) against the false positive rate (1 - specificity) at various classification thresholds. In other words, the model's sensitivity corresponds to the model's ability to detect patients (ENDO+) while the model's specificity corresponds to the model's ability to detect a non-patient (ENDO-). The ROC curve helps assess the model's ability to correctly identify true positives while minimizing false positives.
  The area under the ROC curve (AUC) can be interpreted as the probability that, among two randomly chosen subjects, a patient and a non-patient, the value of the marker is higher for the patient than for the non-sick. An AUC of 0.5 (50%) indicates that the marker is non-informative. An increase in AUC indicates an improvement in discriminatory abilities, with a maximum of 1.0 (100%).
Pelvic pain intensity | t0 : Between the second and the fifth day of the menstrual cycle, before watching an empathy-inducing video
  Pelvic pain will be assessed using a Visual Analogue Scale (VAS). The visual analog scale (VAS) is a validated, unidimensional subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."

OTHER OUTCOMES:
Quality of life (for the ENDO+ group only) | t0 : Between the second and the fifth day of the menstrual cycle, before wathching an empathy-inducing video
  The quality of life of patients with endometriosis is assessed with the Endometriosis Health Profile questionnaire (EHP-30©)
  EHP-30 is a self-administered questionnaire validated in French to assess the effects that endometriosis can have on the quality of life of women. This questionnaire consists of 30 domains grouped into 5 areas:
  Pain (11 items: n° 1 to 11), Control and helplessness (6 items: n°12 to 17), Emotional well-being (6 items: n°18 to 23), Social support (4 items: n°24 to 27), Self-image (3 items: n°28 to 30). Each item is rated on a Likert scale (Never=0, Rarely=1, Sometimes=2, Often=3, Always=4). Each domain is then represented by a score calculated on a scale from 0 (indicating the best possible state of health) to 100 (indicating the worst possible state of health): Domain score = [sum of responses to each item in the domain] / [4 (= maximum item response) × number domain items] × 100
Score of pain (for the ENDO+ group only) | t0 : Between the second and the fifth day of the menstrual cycle, before wathching empathy-inducing video
  The score of pain of patients with endometriosis is assessed with the French version of the Endometriosis Health Profile questionnaire (EHP-30©). The score of the first domain Pain consists of 11 items. Each item is rated on a Likert scale (Never=0, Rarely=1, Sometimes=2, Often=3, Always=4).

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra ALVERGNE, PhD, Study Chair — Centre National de la Recherche Scientifique, France
Locations (1):
- CHU de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No